CLINICAL TRIAL: NCT01385579
Title: A Randomized Controlled Trial of a Direct-to-Patient Outreach Program to Improve Rates of Colorectal Cancer Screening in a Low Income and Racially Diverse Population
Brief Title: Effectiveness of Direct-to-Patient Outreach on Colorectal Cancer Screening Within a Low Income and Diverse Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Bechara Choucair, Adjunct Associate Professor in Family and Community Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU00015652
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-11

CONDITIONS: Malignant Neoplasm of Large Intestine
Keywords: colorectal cancer screening; fecal occult blood testing (FOBT); vulnerable populations; community health center
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care (No Intervention): Patients assigned to the usual care arm may be referred for colorectal cancer screening by their providers per usual health center protocol and practice. They receive no additional outreach by the preventive care care manager.
- Care manager outreach (Experimental): Patients assigned to the intervention arm are mailed a letter informing them that they are due for colorectal cancer screening, educational information about colorectal cancer screening, a fecal occult blood testing (FOBT) kit, and directions on how to complete and return the FOBT kit
  Interventions: Other: Care manager outreach

INTERVENTIONS:
Other: Care manager outreach — Patients assigned to the intervention arm are mailed a letter informing them that they are due for colorectal cancer screening, educational information about colorectal cancer screening, a fecal occult blood testing (FOBT) kit, and directions on how to complete and return the FOBT kit. Patients who do not respond to the mail outreach received up to 3 attempts at telephone outreach by the care manager.
  Arms: Care manager outreach

SUMMARY:
The purpose of this study is to determine if the direct mailing of fecal occult blood testing (FOBT) kits to patients who are due for colorectal cancer screening is an effective way to improve colorectal cancer screening rates within a low income and racially/ethnically diverse population.

DETAILED DESCRIPTION:
Patients ages 50 to 80 who are identified through the electronic health record as not being up to date on colorectal cancer screening are eligible for the study and will be randomly assigned to the intervention or usual care group. Individuals in the intervention group will be mailed a letter informing them that they are due for colorectal cancer screening, educational material regarding colorectal cancer screening, a fecal occult blood testing (FOBT) kit, directions on how to use and return the FOBT kit. The proportion of patients assigned to the intervention versus usual care groups who complete a guideline recommended form of colorectal cancer screening within 4 months of the initiation of outreach will be compared.

ELIGIBILITY:
Inclusion Criteria:

Ages 50 to 80 as of 12/31/2009 At least 2 visits to the community health center between 7/1/2008 and 12/31/2009

Exclusion criteria:

Documented fecal occult blood testing (FOBT) within 1 year (between 1/1/2009 and 12/31/2009) Documented sigmoidoscopy within 5 years (between 1/1/2005 and 12/31/2009) Documented colonoscopy within 10 years (between 1/1/2000 and 12/31/2009)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bechara N Choucair, MD, Principal Investigator — Northwestern University, Feinberg School of Medicine, Department of Family and Community Medicine
Locations (1):
- Heartland International Health Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Jean-Jacques M, Kaleba EO, Gatta JL, Gracia G, Ryan ER, Choucair BN. Program to improve colorectal cancer screening in a low-income, racially diverse population: a randomized controlled trial. Ann Fam Med. 2012 Sep-Oct;10(5):412-7. doi: 10.1370/afm.1381. PMID 22966104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All eligible patients within the health center were randomized to usual care or care manager outreach. Eligibility for randomization was assessed on 12/31/2009. Outreach was conducted from 2/25/2010 through 4/30/2010.
Period: Overall Study
Arm/Group | Usual Care | Care Manager Outreach
Started | 98 | 104
Completed | 98 | 104
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Care Manager Outreach | Total
Number analyzed (Participants) | 98 | 104 | 202
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (8) | 60 (7) | 60 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 67 | 125
  Male | 40 | 37 | 77

OUTCOME MEASURES:

1. Primary Outcome: Completion of a Colorectal Cancer Screening
Description: Patients who have documentation within the electronic health record of completion of a guideline approved form of colorectal cancer screening (colonoscopy, sigmoidoscopy, or fecal occult blood testing (FOBT)) within 4 months of the initiation of the outreach intervention (by June 30, 2010)
Time Frame: within 4 months of the initiation of outreach (by June 30, 2010)
Measure: Number; unit: participants
Arm/Group | Usual Care | Care Manager Outreach
Number analyzed (Participants) | 98 | 104
participants | 5 | 31

ADVERSE EVENTS:
Arm/Group | Usual Care | Care Manager Outreach
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/104
Other Adverse Events (participants affected / at risk) | 0/98 | 0/104

LIMITATIONS AND CAVEATS:
Single site study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No